CLINICAL TRIAL: NCT01022450
Title: Rhabdomyolysis - A Retrospective Study in Hospitalized Patients
Brief Title: Study of the Causes of the Breakdown of Muscle Fibers in Hospitalized Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Fe-Lin Lin Wu / Associate Professor, Director, Graduate Institute of Clinical Pharmacy, College of Medicine, National Taiwan University
Other Study IDs: 200911033R
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Rhabdomyolysis; Myopathy; Acute Renal Failure; Neuroleptic Malignant Syndrome
Keywords: rhabdomyolysis; myopathy; acute renal failure; neuroleptic malignant syndrome; Pharmaceutical Preparations; Hydroxymethylglutaryl-CoA Reductase Inhibitors; fibrates; creatine kinase
MeSH Terms: conditions — Rhabdomyolysis; Muscular Diseases; Acute Kidney Injury; Neuroleptic Malignant Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. Analyze the various causes of breakdown of muscle fibers in hospitalized patients.
2. Analyze the characteristics of these patients in Taiwan (including the drugs history, risk factors and the incidence of complications).

DETAILED DESCRIPTION:
1. Find the causes of breakdown of muscle fibers in hospitalized patients through medical record review.

   * especially drug-related
2. Find the risk factors of muscle fibers breakdown.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to The National Taiwan University Hospital during 2003/1/1~2008/12/31 with the following discharge diagnosis: myoglobinuria, rhabdomyolysis, myopathy, toxic myopathy, malignant hyperthermia, neuroleptic malignant syndrome, polymyositis, myalgia and had acute neuromuscular illness presentations and serum creatinine kinase (CK) more than 5 times the upper limit of normal (male > 900 IU/L; female > 835 IU/L).

Exclusion Criteria:

* Patients with recent myocardial infarction or stroke, unless clinical history, examination, or electromyography showed a concomitant myopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who admitted to The National Taiwan University Hospital during 2003/1/1~2008/12/31 with rhabdomyolysis or related muscle diseases dignosis and clinical presentation.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fe-Lin L Wu, MSCP, PhD, Principal Investigator — Graduate Institute of Clinical Pharmacy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan